CLINICAL TRIAL: NCT01421251
Title: The Safety of GSK Biological's H1N1 Pandemic Vaccine in Manitoba, Canada
Brief Title: H1N1 Vaccine Safety in Manitoba, Canada
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: International Centre for Infectious Diseases, Canada (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: ICID-2011-H1N1-01
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: H1N1 Influenza
Keywords: H1N1; Flu; Influenza; Vaccine; Manitoba; Canada; Safety
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — None collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Matched cohorts - population based: Two cohorts: vaccinated individuals are matched to unvaccinated individuals on the basis of age, sex, and postal code of residence.

SUMMARY:
Many people worldwide received the monovalent adjuvanted H1N1 vaccine. However, very little is known about the safety of the vaccine, particularly beyond the first few weeks after vaccination. This study will combine data from a well-established immunization registry in Manitoba with data from hospitalization and physician records, to examine the safety of the vaccine in the six month period post-vaccination. Studies on vaccine safety are important as the public's perception of the safety of a vaccine has a major role in its uptake.

DETAILED DESCRIPTION:
The objective of this study is to examine the safety of the H1N1 vaccine administered in Manitoba during the second wave of the pandemic (Oct 2009-Mar 2010) by describing the age sex specific and age standardized incidence rates of certain vaccination adverse events in the vaccinated populations during the first 6 months of follow-up and to compare the rates with those in the non-vaccinated population and the general Manitoba population.

Study design The proposed study will be a retrospective analysis of population based cohorts of subjects whose vaccination status and health events before and after H1N1 vaccination are recorded in various Manitoba databases. All H1N1 vaccinated and unvaccinated individuals are eligible to be included in the study population. There will be no exclusion criteria. The list of specific adverse events of special interest (AESIs) includes: anaphylaxis, Bell's palsy, convulsions, demyelination, encephalitis, Guillain-Barré syndrome, neuritis, vasculitis and various pregnancy outcomes.

Vaccinated individuals will be identified using the Manitoba Immunization Monitoring System (MIMS). Unvaccinated individuals will be identified using the Population Registry. AESIs and other clinically relevant information will be determined using hospital, physician claim and DPIN databases.

The primary statistical analysis will be a comparison of the overall and age specific rates of deaths and AESIs in the vaccinated cohort relative to the non-vaccinated cohort. The two cohorts will be matched on age (month and year of birth), sex and postal code of residence. The analyses will be stratified by specific subgroups: (e.g. pregnant women, persons who are immune suppressed or with autoimmune disorders).

The observed number of events will be determined from the date of first vaccination for each subject and the matched control until the first occurrence of a specific event. Information on events for each person will be derived from the medical claims and hospitalization databases. The person years at risk will be calculated from the date of first vaccination until the first occurrence of the specific event, emigration from Manitoba, or until 6 months after vaccination. Incidence rate ratios and 95% confidence intervals will be calculated by comparing the standardized incidence rates in the vaccinated cohort with those in the matched non vaccinated cohort.

In addition, the observed number of deaths and AESIs in the total vaccinated population and in specific subgroups (as above) will be compared to the expected numbers based on the age sex specific rates in the general Manitoba population. Similar to the matched cohort component, the observed number of events will be determined for the vaccinated individuals from the date of first vaccination until the first occurrence of a specific event, and the person years at risk will be calculated from the date of first vaccination until the first occurrence of the specific event, emigration from Manitoba, or until 6 months after vaccination. The background rate of targeted events will be calculated utilizing information from the mortality, physician claims and hospitalization databases for the total population in Manitoba for the period 2004 2008. Since the risk of some of the events is low, calculating the age sex specific rates based on five years of data will increase the stability of the rates. The expected number of events will be calculated by multiplying the person years at risk by the age sex specific background rate of each targeted event. Standardized incidence ratios (SIRs) or mortality ratios (SMRs) will be calculated as the number of observed events over the number of expected events, with 95% confidence intervals. To assess the absolute burden of an eventual excess in observed number of events the absolute difference between the observed and expected number of events for certain AESIs will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* All 6-month or older Manitoba residents are eligible

Exclusion Criteria:

* None

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of the Province of Manitoba, population approximately 1.2 million
Sampling Method: Non-Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Effects of H1N1 vaccination | One year
  Incidence rate ratios of certain vaccination adverse effects

SECONDARY OUTCOMES:
Incidence Ratios of Adverse Effects | One year
  Standardized incidence ratios of certain adverse events in relation to history of H1N1 vaccination.
Sex-specific adverse effects of vaccination | One year
  Determination of sex-specific adverse effects following H1N1 vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Mahmud, M.D., Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- International Centre for Infectious Diseases, Winnipeg, Manitoba, Canada